CLINICAL TRIAL: NCT04303403
Title: Phase Ib Study Evaluating Safety and Tolerability of Combination Trametinib and Ruxolitinib in Patients With Advanced RAS Mutant Colorectal Cancer and Pancreatic Adenocarcinoma
Brief Title: Study of Trametinib and Ruxolitinib in Colorectal Cancer and Pancreatic Adenocarcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CTMT212XSG01T
Record Dates: First submitted 2018-09-25; First posted 2020-03-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Colorectal Cancer; Pancreatic Adenocarcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — trametinib; ruxolitinib

STUDY DESIGN:
Intervention Model Description: The first part of this study will be a standard 3+3 dose-escalating
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose Escalation and Expansion (Experimental): Dose Escalation:
  Trametinib 2mg daily monotherapy for 14 days. Followed by combination oral trametinb (2mg starting dose) daily and oral ruxolitinib (5mg starting dose) twice daily at assigned doses.
  Dose Expansion:
  Combination oral trametinb daily and oral ruxolitinib twice daily at the maximum tolerated dose (MTD) established at the Dose Escalation phase.
  A cycle of therapy will comprise of 28 days of combination trametinib and ruxolitinib treatment.
  Interventions: Drug: Trametinib; Drug: Ruxolitinib

INTERVENTIONS:
Drug: Trametinib — Taken orally once daily
  Other Names: Mekinist
Drug: Ruxolitinib — Taken orally twice daily
  Other Names: Jakafi

SUMMARY:
The purpose of this research study to find out if the drug trametinib in combination with ruxolitinib is safe, tolerable and has beneficial effects in people who has certain type of cancers including the type that you have. Patients with RAS mutant colorectal cancer and pancreatic adenocarcinoma are invited to participate in this study. This is the first time that both trametinib and ruxolitinib are studied in combination. Trametinib is marketed in several countries with the brand name Mekinist® for the treatment of melanoma (a type of skin cancer). Trametinib has been studied extensively in cancer and has been tested in many patients. Ruxolitinib is an oral inhibitor of JAK1 and JAK2 tyrosine kinases and is approved for treatment of adult polycythemia vera and myelofibrosis. Ruxolitinib has been studied extensively in many patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients (male or female) ≥ 21.
* Patients with histological diagnosis of RAS mutant advanced colorectal and pancreatic adenocarcinoma having received at least 1 prior line of systemic therapy. Pancreatic cancer patients with KRAS mutation detected on plasma profiling having received at least 1 prior line of systemic therapy.
* Patients must have at least one measurable lesion according to Response Evaluation Criteria in Solid Tumours (RECIST) criteria version 1.1.
* Life expectancy of at least 3 months.
* Written informed consent that is consistent with ICH-GCP guidelines.
* Eastern Cooperative Oncology Group (ECOG) performance score ≤ 2.
* Have adequate organ and hematologic function, as determined by:

  * Absolute neutrophil count (ANC) ≥ 1,500/μl.
  * Platelets ≥ 100,000/μl.
  * Haemoglobin ≥ 9g/dL.
  * Aspartate Amino Transferase (AST)/ Alanine Amino Transferase (ALT) ≤ 2.5 x upper limit of normal (ULN ≤ 5 x ULN is acceptable if liver metastases are present).
  * Total bilirubin ≤1.5 x ULN (< 3 ULN for patients with Gilbert syndrome).
  * Creatinine clearance ≥ 60ml/min.
  * Prothrombin time and activated partial thromboplastin time ≤ 1.5 x upper limit of normal (ULN) per institutional laboratory normal range.
  * Ejection fraction ≥ 50% with no symptoms attributable to heart failure.
* Have normal QT interval on screening electrocardiogram (ECG) evaluation, defined as QT interval corrected (Fridericia) (QTcF) of ≤450 ms in males or ≤470 ms in females.
* For female patients of childbearing potential, a negative pregnancy test must be documented prior to enrolment.
* Female and male patients who are fertile must agree to use a highly effective form of contraception with their sexual partners throughout study participation.
* Have the willingness and ability to comply with scheduled visits and study procedures.

Exclusion Criteria:

* Received cytotoxic chemotherapy, investigational agents, or radiation within 14 days of study drug commencement, or 5 half-lives, whichever is shorter, and with recovery of clinically significant toxicities from that therapy.
* Received monoclonal antibodies or had surgery within 30 days of the first dose of study drug.
* Have been diagnosed with another primary malignancy within the past 3 years of study drug commencement (except for adequately treated non-melanoma skin cancer, cervical cancer in situ, or prostate cancer).
* Have CNS metastases that are symptomatic, neurologically unstable, or requiring an increasing dose of corticosteroids.
* Have meningeal involvement or spinal cord compression.
* Have significant, uncontrolled, or active cardiovascular disease, specifically including, but not restricted to:

  * Myocardial infarction (MI) within 6 months prior to the first dose.
  * Unstable angina within 6 months prior to first dose.
  * History of congestive heart failure (CHF).
  * History of clinically significant atrial arrhythmia.
  * Any history of ventricular arrhythmia.
  * Cerebrovascular accident or transient ischemic attack within 6 months prior to first dose.
* Have history or the presence of pulmonary interstitial disease or drug related pneumonitis.
* Have an ongoing or active infection.
* Patients with active HBV and HCV are excluded unless they are undergoing treatment for HBV and HCV.
* Have a history of or active significant gastrointestinal (GI) bleeding within 3 months of the first dose.
* Patients who are on immunosuppressive therapy.
* Patients who have retinal vein occlusion and retinal pigment epithelial detachment.
* On medications which are potent and moderate inhibitor and inducers of CYP3A4.
* Patients with moderate to severe hepatic impairment (Child Pugh B and C).
* Patients with history of severe allergic skin reactions or current skin conditions.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2018-07-31 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 28 days (1 cycle)
  Highest dose level at which less than one-third of the patients in the dose level experienced dose limiting toxicities (DLTs) during the first cycle of treatment

SECONDARY OUTCOMES:
Frequency and severity of treatment-emergent Adverse Events and Serious Adverse Events | From time of first study drug administration until 30 days after last dose of study drug
  To assess the safety of the drug combination. During the dose escalation phase, this includes the incidences of dose limiting toxicities during the first 2 cycles of treatment.
Changes between baseline and post-baseline hematology laboratory parameters during treatment - Haemoglobin | From time of first study drug administration until 30 days after last dose of study drug
  Unit of measure: g/dL. To assess the safety of the drug combination
Changes between baseline and post-baseline hematology laboratory parameters during treatment - White blood count, Platelets, Absolute neutrophil count | From time of first study drug administration until 30 days after last dose of study drug
  Unit of measure: x 10^9/L. To assess the safety of the drug combination.
Changes between baseline and post-baseline hematology laboratory parameters during treatment - Neutrophils | From time of first study drug administration until 30 days after last dose of study drug
  Unit of measure: Percentage component of white blood cells. To assess the safety of the drug combination.
Changes between baseline and post-baseline biochemistry laboratory parameters during treatment - Urea, Sodium, Potassium, Chloride, Bicarbonate, Glucose, Magnesium, Calcium, Phosphate, Total cholesterol, High and low density lipoprotein, Triglycerides | From time of first study drug administration until 30 days after last dose of study drug
  Unit of measure: mmol/L. To assess the safety of the drug combination
Changes between baseline and post-baseline biochemistry laboratory parameters during treatment - Uric acid, Creatinine, Total bilirubin | From time of first study drug administration until 30 days after last dose of study drug
  Unit of measure: umol/L. To assess the safety of the drug combination
Changes between baseline and post-baseline biochemistry laboratory parameters during treatment - Total protein, Albumin | From time of first study drug administration until 30 days after last dose of study drug
  Unit of measure: g/L. To assess the safety of the drug combination
Changes between baseline and post-baseline biochemistry laboratory parameters during treatment - Alkaline phosphatase, Alanine transaminase, Aspartate transaminase, Lactate dehydrogenase, Beta-human chorionic gonadotrophin | From time of first study drug administration until 30 days after last dose of study drug
  Unit of measure: U/L. To assess the safety of the drug combination
Frequency of dose interruptions | From time of first study drug administration until 30 days after last dose of study drug
  To assess the tolerability of the drug combination.
Frequency of dose reductions | From time of first study drug administration until 30 days after last dose of study drug
  To assess the tolerability of the drug combination
Pharmacokinetics (PK): Trough concentrations of trametinb | From cycle 1-6 of study (each cycle is 28 days)
  Trough concentrations of trametinb at different cycles of combination treatment with ruxolitinib
Tumour Markers: CEA and CA 19-9 in blood samples | From cycle 1 up to last cycle of treatment (each cycle is 28 days)
  Changes from baseline tumour markers (CEA and CA 19-9) in blood samples
Overall Response Rate | From time of first study drug administration until first occurrence of disease progression, up to 2 years
  The best overall response is the best response recorded from the start of the treatment until disease progression (PD)/ recurrence (taking as reference for PD the smallest measurements recorded since the treatment started).
Disease Control Rate | From time of first study drug administration until best overall response, first occurence of disease progression, up to 2 years
  Percentage of patients who have achieved complete response, partial response and stable disease in accordance to RECIST 1.1.
Progression Free Survival | From time of first study drug administration until first occurence of disease progression, or death from any cause, up to 2 years
  Time elapsed between treatment initiation and tumour progression or death from any cause, with censoring of patients who are lost to follow-up.
Overall Survival | From time of first study drug administration to death from any cause, up to 2 years
  Time elapsed between treatment initiation and death from any cause, with censoring of patients who are lost to follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: David Tai, MD, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No